CLINICAL TRIAL: NCT04031898
Title: Real World Treatment Patterns, Clinical Outcomes and EGFR / T790M Testing Practices in EGFR-Mutated Advanced Non-Small Cell Lung Cancer Patients Receiving First-Line TKI Therapy
Brief Title: Treatment Patterns, Outcomes and Testing in EGFRm NSCLC Patients With EGFR TKI 1L Across Europe (REFLECT)
Acronym: REFLECT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5162R00009
Record Dates: First submitted 2019-07-04; First posted 2019-07-24 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Lung Cancer
Keywords: EGFR TKI; retrospective; treatment patterns; real world evidence
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- full analysis set: All eligible patients who meet all inclusion criteria and none of the exclusion criteria
  Interventions: Other: Non Interventional

INTERVENTIONS:
Other: Non Interventional — This is a non interventional, observational, retrospective study including patients with EGFR-mutated advanced NSCLC, treated with 1st or 2nd generation EGFR TKI therapy in first line

SUMMARY:
Multinational, multi-center medical record review to describe the treatment patterns, clinical outcomes, and EGFR / T790M testing practices in EGFR-mutated advanced NSCLC patients receiving first-line EGFR TKI therapy in Europe.

DETAILED DESCRIPTION:
The aim is to generate real-life data on treatment patterns of the EGFR-mutated advanced NSCLC patients receiving first- or second-generation EGFR TKI in first line of therapy as provided per routine practice in eight countries. An approximate number of 820 patients will take part in the REFLECT study.

It is anticipated that data, generated from the proposed large cohort across centers in Europe, will facilitate a better understanding of unmet medical needs in first line of treatment and will provide a platform for improving patients' management.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of locally advanced unresectable or metastatic NSCLC;
* Aged at least 18 years at first diagnosis of locally advanced/metastatic NSCLC;
* Lab-confirmed EGFR mutation;
* Received a first- or second-generation EGFR TKI as first-line treatment for advanced/metastatic disease;
* First-line EGFR TKI (afatinib, gefitinib, erlotinib) initiated between January 1, 2015 and June 30, 2018;
* Patients may be alive or deceased at the time of medical record review.

Exclusion Criteria:

* Patients enrolled at any time in an interventional clinical trial for an experimental treatment related to EGFR-mutated NSCLC;
* Patients receiving any systemic therapy for locally advanced or metastatic NSCLC prior to first-line EGFR TKI treatment in the locally advanced/metastatic setting;
* Missing or unknown data on any of the following key study dates:

  * Date of initial NSCLC diagnosis;
  * Date of first diagnosis of or progression to advanced/metastatic NSCLC;
  * Date of first-line EGFR TKI initiation for advanced/metastatic disease;
  * Date of death or last available follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: EGFR-Mutated Advanced Non-Small- cell Lung Cancer Patients Receiving First-Line EGFR TKI Therapy
Sampling Method: Non-Probability Sample
Enrollment: 896 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
First- or second-generation EGFR TKI used in first-line therapy | From date of initiating EGFR TKI in first line until the end of available follow-up or death, if this occurs before; assessed up to 60 months
  Frequency distribution of first-line EGFR TKI of first- or second generation prescribed: erlotinib, gefitinib, or afatinib
Proportion of patients progressing on first line EGFR TKI therapy and describe the time to progression | From date of initiating EGFR TKI in first line until the earliest of progression, death or end of available follow-up, whichever occur first; assessed up to 60 months
  Proportion of patients with a progression event during first-line EGFR TKI therapy or other evidence recorded in the patient's medical records deemed by the clinician to be indicative of progression; Time to progression, defined as time from EGFR TKI therapy initiation in the first-line locally advanced or metastatic setting until the earliest of progression death, or end of available follow-up (i.e., progression-free survival); Proportion of patients discontinuing first-line EGFR therapy for reasons other than progression event or death
Proportion of patients receiving second-line therapy and type of second-line therapy among patients progressing on first line EGFR TKI therapy | From date of initiating EGFR TKI in first line until date of starting second-line therapy; assessed up to 60 months
  Proportion of patients prescribed second-line therapy, as well as time to second-line therapy initiation, as defined by time from first-line EGFR TKI discontinuation until the earliest of second-line initiation, death, or end of available follow-up; Frequency distribution of the second-line therapy regimen (chemotherapy, osimertinib, other EGFR TKI, I/O therapy, or other therapy) among patients initiating second-line therapy.

SECONDARY OUTCOMES:
Patients' demographic and baseline disease characteristics | From date of initial diagnosis of NSCLC or metastatic disease, whichever is diagnosed first until the end of available follow-up or death, if this occurs before; assessed up to 60 months
  Patients' demographics, including: sex (male/female), and age at EGFR TKI initiation.
  Baseline disease characteristics, including:
  Smoking status at initial NSCLC diagnosis, Tumor histology and disease stage at initial NSCLC diagnosis, Eastern Cooperative Oncology Group (ECOG) performance status at initial NSCLC diagnosis and at EGFR TKI initiation, Treatment history: for patients initially diagnosed at earlier-stage disease, cancer-directed and palliative therapies received before first diagnosis of or progression to advanced/metastatic EGFR-mutated NSCLC.
Type of sample & test used to determine the EGFR mutation and type of EGFR mutation identified | From date of metastatic disease diagnostic until the end of available follow-up or death, if this occurs before; assessed up to 60 months
  Molecular testing patterns, including: type of sample/test used to assess the EGFR mutation, for example: primary/secondary tumor, tissue/cytology or blood sample; Molecular testing results: EGFR mutation type (exon 19 deletion, L858R mutation, other).
Proportion of patients with brain metastases (BM) among metastatic patients and the overall survival (OS) expectation in the group of patients with BM | From date of metastatic disease diagnostic until the first BM diagnosis; From first BM diagnosis to the start of first-line EGFR TKI therapy, end of available follow-up or death, if this occurs before; all assessed up to 60 months
  Incidence and time to development of BM from first diagnosis of locally advanced or metastatic NSCLC, including:
  Proportion of patients with BM since diagnostic of metastatic disease and proportion of patients with BM developed during treatment, Type of test used to confirm BM diagnosis (e.g., tissue biopsy, imaging, spinal tap, neurologic exam), Proportion of patients who have BM at start of first-line EGFR TKI therapy. Proportion of patients with no development of BM, Patients' demographic and clinical characteristics associated with development of BM, Incidence of BM and time to development of BM from start of first-line EGFR TKI therapy, Proportion of patients prescribed treatments for BM and type of therapy Overall survival (in months) measured from first diagnosis of BM to the date of death from any cause, with patients last known to be alive censored at the date of last available follow-up.
Proportion of patients with leptomeningeal disease (LM) among metastatic patients and the overall survival (OS) | From date of metastatic disease diagnostic until the LM diagnosis; From LM diagnosis to the start of first-line EGFR TKI therapy, end of available follow-up or death, if this occurs before; all assessed up to 60 months
  Incidence and time to development of LM disease from first diagnosis of locally advanced or metastatic NSCLC, including:
  Proportion of patients with LM at first diagnosis of metastatic disease, Type of test to confirm LM diagnosis (cerebrospinal fluid cytology, tissue, imaging, etc.), Proportion of patients who have LM at start of first-line EGFR TKI therapy, Proportion of patients who later develop (during treatment) LM, Proportion of patients with no development of LM, Incidence of LM and time to development of LM from start of first-line EGFR TKI therapy.
  Overall survival (in months) measured from first diagnosis of LM disease to the date of death from any cause, with patients last known to be alive censored at the date of last available follow-up.
Proportion of patients where the first-line therapy with first- or second-generation EGFR TKI is associated with any other systemic therapy, including the type of systemic therapy | From date of initiating EGFR TKI in first line until the earliest of progression, death or end of available follow-up, whichever occurs first; assessed up to 60 months
  Proportion of patients prescribed other systemic treatments (chemotherapy, osimertinib, other EGFR TKI, I/O therapy, or other therapy) in combination with first-line EGFR TKI therapy.
Proportion of patients tested for T790M mutation and the proportion of patients with positive mutation among patients progressing on first-line EGFR TKI therapy | From date of initiating EGFR TKI in first line until the earliest of progression, death or end of available follow-up, whichever occurs first; assessed up to 60 months
  Proportion of patients tested for T790M mutation and among those tested, the proportion who were positive for the mutation, including:
  Binary distribution of T790M mutation testing and, among those tested, the proportion with a positive result, Type of test used to assess the T790M mutation (tissue/cytology or blood sample).
  Among patients tested and positive for T790M mutation, what proportion receives treatment with osimertinib - applicable study measures include binary distribution of osimertinib treatment initiation, and requency distribution of the line of therapy (second- or later-line in the metastatic setting) in which osimertinib was initiated.
Proportion of patients receiving second-line therapy and type of second line therapy received among patients progressing on first-line EGFR TKI therapy and tested for T790M mutation | From date of initiating second-line therapy until the earliest of progression, death or end of available follow-up, whichever occurs first; assessed up to 55 months
  Among patients progressing on first-line EGFR TKI therapy and tested for T790M, proportion who receive (or not) second-line therapy and the second-line therapy selection (chemotherapy, osimertinib, other EGFR TKI, I/O therapy, or other therapy), including:
  Proportion of patients prescribed second-line therapy, as well as time to second-line therapy initiation, as defined by time from first-line EGFR TKI discontinuation until the earliest of second-line initiation, death, or end of available follow-up, Among patients initiating second-line therapy, frequency distribution of the second-line therapy regimen observed (chemotherapy, osimertinib, other EGFR TKI, I/O therapy, or other therapy).
Proportion of patients receiving second-line therapy and type of second line therapy received among patients progressing on first-line EGFR TKI therapy and not tested for T790M | From date of initiating second-line therapy until the earliest of progression, death or end of available follow-up, whichever occurs first; assessed up to 55 months
  Among patients progressing on first-line EGFR TKI therapy and not tested for T790M, proportion who receive (or not) second-line therapy and the second-line therapy selection (chemotherapy, osimertinib, other EGFR TKI, I/O therapy, or other therapy), including:
  Proportion of patients prescribed second-line therapy, as well as time to second-line therapy initiation, as defined by time from first-line EGFR TKI discontinuation until the earliest of second-line initiation, death, or end of available follow-up, Among patients initiating second-line therapy, frequency distribution of the second-line therapy regimen observed (chemotherapy, osimertinib, other EGFR TKI, I/O therapy, or other therapy).
How the proportion of patients receiving second-line therapy differs between patients tested for T790M mutation and patients not tested for T790M mutations | From date of initiating second-line therapy until the earliest of progression, death or end of available follow-up, whichever occurs first; assessed up to 55 months
  Proportion of patients prescribed second-line therapy, as well as time to second-line therapy initiation, as defined by time from first-line EGFR TKI discontinuation until the earliest of second-line initiation, death, or end of available follow-up among patients tested and not tested for T790M mutation.
Proportion of patients receiving third- or later-line therapy and type of this therapy and to explore whether the proportion receiving third-/later-line therapies varies by the second-line therapy category received | From date of initiating second-line therapy until the earliest of progression, death or end of available follow-up, whichever occurs first; assessed up to 50 months
  Proportion of patients prescribed third- or later lines of therapy and type of therapies selected (chemotherapy, osimertinib, other EGFR TKI, I/O therapy, or other therapy), and how these proportion varies by the second-line therapy category received.
Overall survival (OS) expectation for all patients from first diagnosis of locally advanced or metastatic disease and from start of first-line EGFR TKI therapy | From date of metastatic disease diagnostic or start of first-line EGFR TKI therapy until the end of available follow-up or death, if this occurs before; assessed up to 60 months
  OS (in months) measured overall from first diagnosis of or progression to locally advanced or metastatic disease, OS from start of first-line EGFR TKI therapy to the date of death from any cause, with patients last known to be alive censored at the date of last available follow-up.
Incidence of other mutations, in case additional molecular testing was performed either at the time of initial EGFR testing or at the time of T790M testing | From date of metastatic disease diagnostic until end of available follow-up or death, if this occurs before; assessed up to 60 months
  Proportion of patients with other positive mutations, in case additional molecular testing were performed at the time of initial EGFR testing or at the time of T790M testing (e.g., KRAS, BRAF, ROS1 translocation, PD-L1 expression, MET amplification, ALK rearrangement, RET rearrangement, HER2 exon 20 insertion, TP53, others).

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Syrigos, Prof., Principal Investigator — Oncology Unit, Athens University School of Medicine,
Locations (1):
- Research Site, Wien, Bulgaria

REFERENCES:
- [Derived] Janzic U, Turnsek N, Dediu M, Donev IS, Lupu R, Teodorescu G, Ciuleanu TE, Pluzanski A. Real-World Testing Practices, Treatment Patterns and Clinical Outcomes in Patients from Central Eastern Europe with EGFR-Mutated Advanced Non-Small Cell Lung Cancer: A Retrospective Chart Review Study (REFLECT). Curr Oncol. 2022 Aug 17;29(8):5833-5845. doi: 10.3390/curroncol29080460. PMID 36005198
- [Derived] Lampaki S, Mountzios G, Georgoulias V, Rapti A, Xanthakis I, Baka S, Mavroudis D, Samantas E, Athanasiadis E, Zagouri F, Charpidou A, Somarakis A, Papista C, Nikolaou A, Anastasopoulou E, Paparepa Z, Syrigos KN. Real-world management patterns in EGFR-mutant advanced non-small-cell lung cancer before first-line adoption of osimertinib: the REFLECT study in Greece. Future Oncol. 2022 Sep;18(28):3151-3164. doi: 10.2217/fon-2022-0386. Epub 2022 Aug 5. PMID 35929414
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5162R00009&attachmentIdentifier=ad28088c-367e-4c50-bc02-f0a50b2403ee&fileName=Synopsis_redacted.pdf&versionIdentifier=